CLINICAL TRIAL: NCT03633643
Title: Single-Dose Versus 3-Day Cotrimoxazole Prophylaxis in Transurethral Resection or Greenlight Laser Vaporisation of the Prostate: A Pragmatic, Multicentre Randomised Placebo Controlled Non-Inferiority Trial
Brief Title: Cotrimoxazole Prophylaxis in Transurethral Resection or Greenlight Laser Vaporisation of the Prostate
Acronym: CITrUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-0104; me17Widmer
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Antimicrobial Prophylaxis in Prostate Surgery
Keywords: Greenlight Laser Vaporisation of the Prostate; Transurethral resection of the prostate; Cotrimoxazole Prophylaxis

STUDY DESIGN:
Intervention Model Description: single-dose application of Cotrimoxazole compared to a 3-day application of Cotrimoxazole
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator): Single-dose Trimethoprim (TMP)/sulfamethoxazole (SMX, i.e. Cotrimoxazole) perioperative as two ampoules of TMP/SMX 400/80 mg (Bactrim Inf Konz®) solved in 250 ml sodium chloride short infusion followed by five oral applications of placebo (lactose tablet; Fagron Gesellschaft mit beschränkter Haftung (GmbH) & Co.KG) at the evening of the surgery and thereafter twice daily on day 1 and 2 after surgery while the patient is in hospital.
  Interventions: Drug: oral applications of Placebo
- Group B (Active Comparator): 3-day application with TMP/SMX (i.e. Cotrimoxazole): Preoperatively as two ampoules of TMP/SMX 400/80mg (Bactrim Inf Konz®) solved in 250 ml sodium chloride short infusion, followed by five oral applications of TMP/SMX 800/160 mg (Nopil forte® tablets) at the evening of the surgery and thereafter twice daily on day 1 and 2 after surgery while the patient is in hospital.
  Interventions: Drug: oral applications of TMP/SMX 800/160 mg (Nopil forte® tablets)

INTERVENTIONS:
Drug: oral applications of TMP/SMX 800/160 mg (Nopil forte® tablets) — five oral applications of TMP/SMX 800/160 mg (Nopil forte® tablets) at the evening of the surgery and thereafter twice daily on day
  1 and 2 after surgery while the patient is in hospital.
  Arms: Group B
Drug: oral applications of Placebo — five oral applications of Placebo at the evening of the surgery and thereafter twice daily on day 1 and 2 after surgery while the patient is in hospital.
  Arms: Group A

SUMMARY:
The optimal duration of antimicrobial prophylaxis (study medication Cotrimoxazole (Trimethoprim/Sulfamethoxazole)) in transurethral resection of the prostate and Greenlight Laser vaporisation of the prostate is investigated by comparing a guideline-conform single-dose prophylaxis (intervention) versus usual clinical care (i.e. 3-day prophylaxis; control) for prevention of urinary tract infections.

DETAILED DESCRIPTION:
Increasing antimicrobial resistance rates have a substantial impact on morbidity, mortality and healthcare costs and is particularly prevalent among urological patients due to an overuse of antimicrobial agents for therapeutical and prophylactic indications. Transurethral resection of the prostate is one of the most frequently performed urological procedures in Switzerland and a single-dose of antimicrobial prophylaxis is recommended to reduce postoperative urinary tract infections. For photoselective vaporisation of the prostate with the Greenlight Laser, a similar operative alternative, there are currently no international guidelines for antimicrobial prophylaxis.

The optimal duration of antimicrobial prophylaxis in transurethral resection of the prostate and Greenlight Laser vaporisation of the prostate is investigated by comparing a guideline-conform single-dose prophylaxis (intervention) versus usual clinical care (i.e. 3-day prophylaxis; control) for prevention of urinary tract infections.

The study medication Cotrimoxazole (Trimethoprim/Sulfamethoxazole) is a routinely used antimicrobial substance recommended in international and in-house guidelines for antimicrobial prophylaxis and treatment of urinary tract infections. Perioperative antimicrobial prophylaxis will be Cotrimoxazole short infusion in both groups. Postoperative study medication packages consists of either five tablets of placebo or five tablets of Cotrimoxazole (Nopil forte®) 800/160mg using licensed product repacked in a new immediate container which is blinded

ELIGIBILITY:
Inclusion Criteria:

* Obstructive voiding disorder (e.g. benign prostate hyperplasia, obstructive prostate cancer)
* Planned Transurethral resection of the prostate (TURP) or Greenlight Laser (GL)

Exclusion Criteria:

* Evidence for (catheter associated-) UTI, with or without antibiotic treatment in the last 7 days prior to randomisation.
* Any evidence of a history of positive urine culture (cfu ³105/ml in midstream-urine with no more than two species) and resistance to TMP/SMX in the last 7 days prior to randomisation.
* Known contraindication against study drugs according to the Swissmedic package leaflet (e.g. known liver dysfunction, renal insufficiency; patients with glomerular filtration rate (calculated by the Modification of Diet in Renal Disease (MDRD) or Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) <30ml/min or dialysis patients will be excluded).
* Antibiotic treatment for any reason within 7 days prior to randomisation
* Indication for Antibiotic prophylaxis (AP) for other reasons (e.g. endocarditis prophylaxis, transplanted patients under systemic immunosuppression).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Symptomatic UrinaryTract Infection (UTI) | within 30 days after randomization
  Symptomatic UTI (based on clinical diagnosis) treated with antimicrobial agents

SECONDARY OUTCOMES:
Symptomatic UTI by measured bacteriuria | within 30 days after randomization
  measured bacteriuria of ≥105 cfu/ml treated with antimicrobial agents (key secondary outcome)
Symptomatic cystitis (based on clinical diagnosis) | within 30 days after randomization
  Symptomatic cystitis (based on clinical diagnosis)
Symptomatic epididymitis (based on clinical diagnosis) | within 30 days after randomization
  Symptomatic epididymitis (based on clinical diagnosis)
Symptomatic pyelonephritis (based on clinical diagnosis) | within 30 days after randomization
  Symptomatic pyelonephritis (based on clinical diagnosis)
Symptomatic prostatitis (based on clinical diagnosis) | within 30 days after randomization
  Symptomatic prostatitis (based on clinical diagnosis)
Symptomatic urethritis (based on clinical diagnosis) | within 30 days after randomization
  Symptomatic urethritis (based on clinical diagnosis)
Urosepsis (based on clinical diagnosis) | within 30 days after randomization
  Urosepsis (based on clinical diagnosis)
Prescription of antibiotics (for any reason) | within 30 days after randomization
  Prescription of antibiotics (for any reason)
Prescribed defined daily doses (DDD) of antibiotics (cumulative sum of DDD) day 30) | within 30 days after randomization
  Prescribed defined daily doses (DDD) of antibiotics (cumulative sum of DDD)
Asymptomatic bacteriuria of ≥105 cfu/ml treated with antimicrobial agents | within 30 days after randomization
  Asymptomatic bacteriuria of ≥105 cfu/ml treated with antimicrobial agents
Detection of multidrug-resistant bacteria in Urine culture | within 30 days after randomization
  Detection of multidrug-resistant bacteria in Urine culture
Any Clostridium difficile-associated infection | within 30 days after randomization
  Any Clostridium difficile-associated infection
Duration of catheterisation (cumulative sum of days between randomisation and end of catheterisation or day 30) | within 30 days after randomization
  Duration of catheterisation (cumulative sum of days between randomisation and end of catheterisation or day 30)
Duration of hospital stay (cumulative sum of Hospital days between randomisation and day 30) | within 30 days after randomization
  Duration of hospital stay (cumulative sum of Hospital days between randomisation and day 30)
Duration of intensive care unit (ICU) stay (cumulative sum of ICU days between randomisation and day 30) | within 30 days after randomization
  Duration of intensive care unit stay (cumulative sum of ICU days between randomisation and day 30)
Re-hospitalisation (within 30 days after randomisation) | within 30 days after randomization
  Re-hospitalisation (within 30 days after randomisation)
Change of International Prostate Symptom Score (prior to randomisation and at day 30 after randomisation) | within 30 days after randomization
  Change of International Prostate Symptom Score (prior to randomisation and at day 30 after randomisation)
Change of Quality of life Score (prior to randomisation and at day 30 after randomisation) | within 30 days after randomization
  Change of Quality of life Score (prior to randomisation and at day 30 after randomisation)
All-cause mortality | within 30 days after randomization
  All-cause mortality
Total adverse events | within 30 days after randomization
  Total adverse events
Total serious adverse events | within 30 days after randomization
  Total serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Widmer, Prof.,MD,Dr., Principal Investigator — Division of Infectious Diseases and Hospital Epidemiology
Locations (5):
- Switzerland (5):
  - St. Claraspital, Department of Urology, Basel, Canton of Basel-City
  - Kantonsspital Aarau, Department of Urology, Aarau
  - University Hospital Basel, Division of Infectious Diseases and Hospital Epidemiology, Basel
  - Kantonsspital Baselland, Department of Urology, Liestal
  - University Hospital Zurich, Department of Urology, Zurich

REFERENCES:
- [Derived] Speich B, Bausch K, Roth JA, Hemkens LG, Ewald H, Vogt DR, Bruni N, Deuster S, Seifert HH, Widmer AF. Single-dose versus 3-day cotrimoxazole prophylaxis in transurethral resection or greenlight laser vaporisation of the prostate: study protocol for a multicentre randomised placebo controlled non-inferiority trial (CITrUS trial). Trials. 2019 Feb 19;20(1):142. doi: 10.1186/s13063-019-3237-3. PMID 30782183